CLINICAL TRIAL: NCT05580913
Title: Auto-regulated Resistance-training for Improving Strength in Older Adults
Brief Title: Auto-regulated Resistance-training for Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Phil Chilibeck, Professor, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2972
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Subjective auto-regulation training (Experimental): Participants complete their resistance-training sets to termination based on rating of perceived exertion
  Interventions: Behavioral: Resistance training
- Objective auto-regulation training (Experimental): Participants complete their resistance-training sets to termination based on reaching a critical slow velocity
  Interventions: Behavioral: Resistance training
- Traditional standardized training (Active Comparator): Participants complete their resistance-training sets by lifting a prescribed percentage of their estimated one-repetition maximum (as determined from baseline four-repetition maximum strength testing)
  Interventions: Behavioral: Resistance training

INTERVENTIONS:
Behavioral: Resistance training — 12 weeks of resistance-training performed two times per week

SUMMARY:
This research study is comparing the effect of traditional standardized, subjective auto-regulated, and objective auto-regulated resistance training on physiological adaptations and performance measures in adults aged 50 years or older. Traditional standardized resistance training involves prescribing resistance training as a percentage of an individual's one-repetition maximum (i.e., the maximal weight they can lift one time). Auto-regulated resistance training involves adjusting resistance training based on an individual's performance during the session. Subjective auto-regulation involves the resistance trainee providing a subjective rating of perceived exertion based on repetitions in reserve (on a scale from 1 - 10) to adjust the resistance training prescription. A rating of perceived exertion of 10 would mean that the resistance trainee believes that they have provided maximal effort and believes that they could not have performed an additional repetition during the set nor increased the load. Objective auto-regulation involves adjusting the resistance training prescription from a linear position transducer (a device that has a string that attaches to the barbell and provides a velocity value on each repetition). A slower velocity value means a higher perceived exertion and load used, whereas a faster velocity value means a lower perceived exertion and load used.

DETAILED DESCRIPTION:
Auto-regulated resistance training has emerged as a resistance training paradigm to individualize programming; however, it remains to be elucidated whether auto-regulated resistance training provides a greater benefit than traditional standardized resistance training on physiological adaptations and performance outcomes in older adults. Traditional resistance training involves prescription of intensity as a percentage of the maximal amount of weight an individual can lift (for example, a resistance of 70% of maximal strength is a weight equal to 70% of the maximal weight a person can lift one time. An individual with this prescription would lift this weight for a number of repetitions to failure; i.e. usually 8-10 repetitions). Auto-regulation can be done two ways: "Subjective" auto-regulation involves lifting a weight for a number of repetitions until the individual reaches a certain "rating of perceived exertion". The rating of perceived exertion is on a scale of 1-10, with 10 being the most difficult or maximal exertion. For example, if one was prescribed a rating of perceived exertion of 8 they would lift a weight for a given number of repetitions until they believed they were at an 8/10 on the scale and had 2 repetitions left before failing. "Objective" auto-regulation involves lifting a weight for a given number of repetitions until a predetermined velocity of lifting is reached. For example, once someone starts to get fatigued while performing repeated lifting, the velocity of lifting will slow down. Once they have reached a critical slow velocity, the exercise would be stopped. There is some evidence that auto-regulation improves muscular strength to a greater extent than traditional resistance training in healthy populations.

The research design is a prospective randomized trial comparing three training protocols in 30 participants. Participants will be randomized into one of three groups (n = 10 each), with matching on baseline strength: traditional standardized, subjective auto-regulated, and objective auto-regulated. Training will be twice per week for 12 weeks. Measures include strength assessments, muscle size, and performance of functional tasks.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 50 years of age or greater

Exclusion Criteria:

* Inability to safely perform squat and bench press exercises as determined by the Get Active Questionnaire

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in bench press strength | baseline, 12 weeks
Change from baseline in squat strength | baseline, 12 weeks

SECONDARY OUTCOMES:
Change from baseline in muscle thickness | Baseline, 12 weeks
  Muscle thickness will be determined for the quadriceps, hamstrings, triceps, and pectoralis (males only)
Change from baseline in knee extension strength | Baseline, 12 weeks
Change from baseline for time to sit and stand from a chair five times | Baseline, 12 weeks
Change from baseline in time to complete the "timed up and go" (TUG) test | Baseline, 12 weeks
  Time to stand from a chair, walk around a cone (3 meters) and sit back down in the chair
Change from baseline in time to climb 10 stairs | Baseline, 12 weeks
Change from baseline in time to walk 10 meters | Baseline, 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No